CLINICAL TRIAL: NCT06172244
Title: Acute Effect of Whole Body Vibration on Reaction Speed and Proprioception in the Upper Extremity in Healthy Subjects
Brief Title: Acute Effect of Whole Body Vibration on Reaction Speed and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çağtay Maden (Other)
Responsible Party: Sponsor-Investigator, Çağtay Maden, Assistant professor, Gaziantep Islam Science and Technology University
Organization: Gaziantep Islam Science and Technology University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023/266
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-06

CONDITIONS: Whole Body Vibration
Keywords: whole body vibration; healthy subject; reaction time; proprioception; Upper Extremity

STUDY DESIGN:
Intervention Model Description: A total of 5 sets of vibration will be given at 30 Hz, 2 mm amplitude, 1 minute of application and 1 minute of rest.
Masking Description: In statistical analysis, blinding will be done before and after the application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole body vibration (Experimental): A total of 5 sets of vibration will be given at 30 Hz, 2 mm amplitude, 1 minute of application and 1 minute of rest.
  Interventions: Other: Applying with whole body vibration device

INTERVENTIONS:
Other: Applying with whole body vibration device — A total of 5 sets of vibration will be given at 30 Hz, 2 mm amplitude, 1 minute of application and 1 minute of rest.

SUMMARY:
It will be determined whether the application of whole body vibration has an immediate effect on upper extremity reaction speed and proprioception.

DETAILED DESCRIPTION:
Muscles and tendons are among the mechanisms affected by whole body vibration. In this way, it is thought that TVV indirectly affects the reaction speed of individuals. In the light of this information, this study was planned to investigate how whole body vibration application affects proprioception and reaction speed. The reaction rate and instantaneous effect of the virion given at 30 Hz and 2 mm amplitude in the push-up position on proprioception will be investigated. The aim of this study is to investigate the instantaneous effect of whole body vibration on reaction speed and proprioception in the upper extremity in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18-25
* Those who do not have any orthopedic problems in the upper extremity
* Individuals without any neurological problems
* Those who volunteer to participate in the study

Exclusion Criteria:

* Those who have vertigo

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Nelson Hand Reaction Test | All measurements take 30 minutes for each individual, before and immediately after the application on the same day.
  The participant is asked to sit in the chair with the forearm and hand comfortably resting on the table. The tips of the thumb and index finger are positioned 8-10 cm away from the table, with the tops of the thumb and index finger parallel to each other. The tester asks the individual to hold the ruler between his thumb and index finger. At the same time, the patient is asked to look directly at the middle point of the ruler while holding it between his fingers. As soon as the ruler is released, the person is told to catch the ruler with his thumb and forefinger. The ruler is left and the numerical value on the upper edge of the subject's thumb, where the subject grasps the ruler, is read and recorded.
Reaction Rate Evaluation with Sway Medical Smartphone Application | All measurements take 30 minutes for each individual, before and immediately after the application on the same day.
  The person will sit comfortably on a chair and hold the smartphone with the thumbs on both sides. When the orange screen appears, the phone should quickly rotate the screen in the desired direction. Once you will do the test to learn the application. Then, the application is made three times and the reaction rate is calculated by taking the average time of these three applications.
Upper extremity proprioception measurement | All measurements take 30 minutes for each individual, before and immediately after the application on the same day.
  Elbow flexion, shoulder flexion and abduction 30 and 60 degree angles were measured with a digital goniometer. The elbow and shoulder positions were brought to the desired angle and they were asked to return to the same angle. The angle of deviation was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Çağtay MADEN, Principal Investigator — Gaziantep İslamic Science and Technology University
Locations (1):
- Gaziantep İslamic Science and Technology University, Gaziantep, Şahinbey, Turkey (Türkiye)